CLINICAL TRIAL: NCT06449248
Title: Oral Lichen Planus and Systemical Oncological Comorbidities: Case-control Multicenter Observational Clinical Study
Brief Title: Oral Lichen Planus and Systemical Oncological Comorbidities
Status: Completed | Type: Observational
Sponsor: Catholic University of the Sacred Heart (Other)
Responsible Party: Principal Investigator, Carlo Lajolo, Associate Professor, Catholic University of the Sacred Heart
Other Study IDs: Lichen-Cancer
Record Dates: First submitted 2024-06-03; First posted 2024-06-07 (Actual); Last update posted 2024-06-07 (Actual); Status verified 2024-06

CONDITIONS: Oral Lichen Planus
Keywords: Oral Lichen Planus; Cancer; Retrospective; Multicenter
MeSH Terms: conditions — Lichen Planus, Oral; Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Case Group: 1. Patients of both sexes, consecutively enrolled in a 1:2 ratio
  2. Age over 18 yo
  3. Previous clinical and histological diagnosis of OLP
  Interventions: Other: Checking of appropriateness of OLP diagnosis
- Control Group: 1. Patients of both sexes, consecutively enrolled in a 1:2 ratio
  2. Age over 18 yo

INTERVENTIONS:
Other: Checking of appropriateness of OLP diagnosis — The above mentioned interventions will be carried out through the accurate analysis of patients' clinical records
  Other Names: Checking the presence of any tumor in any body district
  Groups: Case Group

SUMMARY:
Lichen planus (LP) is a chronic mucocutaneous inflammatory disease of unknown etiology.

In its oral variant, oral lichen planus (OLP) has a reported prevalence ranging from 0.5% to 2.2% in the general population. The disease typically occurs between the ages of 30 and 60. Although the pathogenetic mechanism and the triggering factor remain unknown, an immune-mediated pathogenesis and the role of factors such as stress, anxiety, diabetes, other autoimmune diseases, hypertension, intestinal pathologies, chronic liver diseases, hypercholesterolemia, infections have been hypothesized , contact with dental materials, tumors and genetic predisposition to cancer.

Oral lichen planus is one of the potentially malignant disorders, showing a malignant transformation rate of 1.4%.

A preliminary analysis conducted in our research center has shown a correlation between OLP and systemic tumors, both solid and haematological, involving areas not involved in lesions attributable to OLP.

According to these data, the objective of the study is to evaluate whether there is an association between OLP and peripheral tumors, both solid and haematological.

The primary objective will be to investigate the possible existence of a statistically significant association between OLP and the development of systemic oncological pathologies.

Secondary objective will be to investigate the existence of an association between the various forms of OLP and specific oncological pathologies and to evaluate whether the presence of other systemic pathologies and lifestyle factors (diabetes, hypertension, chronic liver disease, smoking, alcohol, infection by HPV, HCV, etc ...) could influence such association (primary outcome).

The objectives will be pursued through the analysis of data collected from the medical records of patients belonging to the General Dentistry and Orthodontic Outpatient Clinics at the "Agostino Gemelli" Teaching Hospital and in the Oral Pathology Outpatient Clinics of the other centers involved.

DETAILED DESCRIPTION:
Lichen planus (LP) is a chronic mucocutaneous inflammatory disease of unknown etiology.

In its oral variant, oral lichen planus (OLP) has a reported prevalence ranging from 0.5% to 2.2% in the general population. The disease typically occurs between the ages of 30 and 60. Although the pathogenetic mechanism and the triggering factor remain unknown, an immune-mediated pathogenesis has been hypothesized and the role of some factors such as stress, anxiety, diabetes, other autoimmune diseases, hypertension, intestinal diseases, chronic liver diseases, hypercholesterolemia, infections, contact with dental materials, tumors and genetic predisposition to cancer.

Oral lichen planus typically has six clinical forms, classified as reticular, erosive, atrophic, plaque, papular, and bullous. The various forms can coexist in a single patient and/or can change over time.

About two-thirds of patients with OLP report oral symptoms that can range from burning to pain. Oral pain is associated in most cases with atrophic or erosive lesions, while other oral symptoms such as burning, xerostomia, and altered taste may be exacerbated by changes in the oral mucosal surface at the lesions' site.

Oral lesions can persist for many years and symptoms and are characterized by periods of quiescence and exacerbation, generally associated with an increase in erythematous and/or ulcerative lesions with consequent pain and hypersensitivity. Patients with quiescent forms, predominantly keratotic and plaque, are generally asymptomatic.

Corticosteroids, applied topically to lesions or administered systemically, are the most widely used group of drugs. The reason for their use is the ability to modulate inflammation and the immune response.

Forms that do not respond to corticosteroid therapy can be treated with immunosuppressive drugs, such as cyclosporine.

The use of antifungals in association with corticosteroid treatment allows for an improvement in the lesions, if they were already overinfected by C. Albicans, and prevents excessive proliferation that could result from the use of corticosteroids.

OLP is one of the potentially malignant disorders, showing a malignant transformation rate of 1.4%.

It is now known that lesions ascribable to OLP, as an expression of a potentially malignant disorder, can turn into neoplasms over time.

A preliminary analysis conducted in our research center has shown a correlation between OLP and systemic tumors, both solid and haematological, involving areas not involved in lesions attributable to OLP.

According to this evidence, the aim of the study is to assess whether there is an association between OLP and distant tumors, both solid and haematological.

The primary objective will be to investigate the possible existence of a statistically significant association between OLP and the development of systemic oncological pathologies. This analysis will be performed on a group of patients affected by OLP compared with a group of patients without OLP.

Secondary objective will be to investigate the possible existence of an association between the different clinical forms of OLP and specific oncological pathologies; furthermore, additional secondary objectives will be to investigate whether the association between OLP and systemic tumors can be influenced by lifestyle factors, such as smoking and alcohol use, and/or by the presence of other systemic diseases (diabetes, hypertension, chronic liver disease , smoking, alcohol, HPV, HCV infection, etc.) The objectives will be pursued through the analysis of data collected from the medical records of patients belonging to the General Dentistry and Orthodontic Outpatient Clinics at the "Agostino Gemelli" Teaching Hospital and in the Oral Pathology Outpatient Clinics of the other centers involved.

ELIGIBILITY:
Inclusion Criteria (Study Group):

1. Patients of both sexes, consecutively enrolled in a 1:2 ratio
2. Age over 18 yo
3. Previous clinical and histological diagnosis of OLP

Exclusion Criteria (Study Group):

1. Age under 18 yo

Inclusion Criteria (Control Group):

1. Patients of both sexes, consecutively enrolled in a 1:2 ratio
2. Age over 18 yo

Exclusion Criteria (Control Group):

1. Age under 18 yo
2. Previous clinical and histological diagnosis of OLP

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study will enroll patients previously treated at the General Dentistry and Orthodontic Outpatient Clinics of the promoter center ("Agostino Gemelli" Teaching Hospital) and associated centers.
Sampling Method: Non-Probability Sample
Enrollment: 1517 (Actual)
Dates: Start 2023-01-02 (Actual); Primary Completion 2023-10-02 (Actual); Study Completion 2023-12-02 (Actual)

PRIMARY OUTCOMES:
Presence of any other tumor | After the enrollment phase (during the subsequent month)
  Researchers will check patient's clinical records looking for any type of tumor

SECONDARY OUTCOMES:
OLP Form and systemic cancer | After the enrollment phase (during the subsequent six months)
  Evaluation of the association between a specific OLP clinical form and the development of systemic cancers
Lifestyle habits and/or infections and systemic tumors | After the enrollment phase (during the subsequent six months)
  Evaluation of the association between specific lifestyle factors and/or infections and the development of systemic cancers

CONTACTS AND LOCATIONS:
Overall Officials: Romeo Patini, Univ. Res., Study Chair — Catholic University of Sacred Heart - Rome
Locations (1):
- Catholic University of Sacred Heart, Roma, Italy

IPD SHARING:
Plan to Share IPD: Yes
Study Design will be shared with other centers participating to the study.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available from the beginning of the enrollment phase until the end of the study.
Access Criteria: Upon request to the PI

REFERENCES:
- [Derived] Gioco G, Schiavelli A, Majorana A, Bardellini E, Abati S, Sardella A, Spadari F, Pellegrini M, Lauritano D, Borgia R, Pentenero M, Sutera S, Arduino PG, Gambino A, Broccoletti R, Biasotto M, Ottaviani G, Azzi L, D'Aiuto A, Gissi DB, Gabusi A, Santarelli A, Mascitti M, Vescovi P, Bortolotti G, Manfredi M, Meleti M, Zino G, Romeo U, Tenore G, Favia G, Limongelli L, Petruzzi M, Dimilito F, Lo Muzio L, Bizzoca ME, Campisi G, Panzarella V, Leuci S, Serpico R, Lucchese A, Colella G, Oteri G, Marciano A, Isola G, Polizzi A, Giudice A, Calabria E, Mariani U, Adamo D, Canfora F, Graziani F, Nisi M, Giuliani M, Ritrovato L, De Micheli F, Rupe C, Scilla F, Patini R, Cordaro M, Mignogna MD, Lajolo C; SIPMO (Italian Society of Oral Pathology and Medicine). Association Between Oral Lichen Planus and Non-Oral Cancers: A Multicentre Case-Control SIPMO Study. Oral Dis. 2025 Nov 24. doi: 10.1111/odi.70152. Online ahead of print. PMID 41286554